CLINICAL TRIAL: NCT01143480
Title: Study of the Effect of Innate Immunity on the Inflammatory Response to Endotoxin
Brief Title: Study of the Effect of Innate on the Inflammatory Response to Endotoxin
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100129; 10-E-0129
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-05-02

CONDITIONS: Asthma; Atherosclerosis; Metabolic Syndrome; Insulin Resistance; Cancer
Keywords: Endotoxin; Innate Immunity; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Asthma; Atherosclerosis; Metabolic Syndrome; Insulin Resistance; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- ABCA1: SNP or allele of interest
- APOE: SNP or allele of interest
- APOL1: SNP or allele of interest
- CD14: SNP or allele of interest
- CD44: SNP or allele of interest
- IRGM: SNP or allele of interest
- ITIH3: SNP or allele of interest
- ITIH4: SNP or allele of interest
- MyD88: SNP or allele of interest
- TIRAP: SNP or allele of interest
- TLR4: SNP or allele of interest
- TLR5: SNP or allele of interest
- TNFa: SNP or allele of interest

SUMMARY:
Background:

- Innate immunity is the process by which white blood cells and other parts of the immune system sense and respond to potential infections by causing an inflammation. Researchers are interested in studying how the body responds to certain environmental factors, and whether the body s response can contribute to chronic illnesses or diseases such as asthma and certain types of cancers.

Objectives:

- To examine how specific genes and proteins in blood cells respond to environmental exposures.

Eligibility:

- Healthy volunteers between 18 and 45 years of age.

Design:

* The study will involve one visit of 45 to 60 minutes.
* Participants will be screened with a brief physical examination and finger stick to determine if they are eligible to donate blood for the study, and will complete a questionnaire about any medications or other drugs (e.g., cigarettes) they may be taking.
* Participants will provide a blood sample for research purposes.

DETAILED DESCRIPTION:
This research study will examine the role of innate immunity on the Inflammatory response of monocytes and macrophages to endotoxin. Approximately 1450 healthy participants aged 18 years and older will be identified and recruited from the Environmental Polymorphism Registry (EPR). The EPR is a long-term project to collect and store up to 15,000 DNA samples for use in research studies from individuals in the greater North Carolina Triangle Region. It is anticipated that approximately 50% of the participants contacted will enroll and about 15% of participants enrolled will withdraw.

This controlled, observational gene association study will recruit participants on the basis of genotype and then observe the phenotype of each participant. There are several SNPs of interest in the genes TIRAP, MyD88, ABCA1, CD14, CD44, ITIH3, ITIH4, TLR4, TNFa, TLR5, IRGM, and APOL1. In addition there are alleles of interest in the gene ApoE. These alleles taken together are considered a polymorphism. For each polymorphism of interest a separate group of participants will be recruited (including heterozygous and homozygous for both the minor and major alleles for each SNP). A maximum of 200 mLs of blood will be obtained from each participant during one visit lasting approximately 1-1.5 hours. Blood monocytes will be isolated from the donated blood samples and cultured to obtain macrophages. The macrophages will be exposed ex vivo to an endotoxin (LPS) and to PAM3CSK4 to determine cell response depending on genotype. In studies of APOL1, a urine specimen will also be collected to evaluate for protein filtration.

The primary objective is to determine associations between select polymorphisms in genes [TIRAP (TIR Associated Protein), MyD88 (Myeloid Differentiation Primary Response Protein 88), ApoE (Apolipoprotein E), ABCA1 (ATP Binding Cassette Transporter A1), CD14, CD44, ITIH3, ITIH4, TLR4, TNFa, TLR5, IRGM, and APOL1] and quantitative in vitro inflammatory functions of two cell types, the macrophage and neutrophil. The primary endpoints of this study for both cell types will be levels of 6 cytokines TNF alpha, IL-6, MIP-2, IL-8, MCP-1, and IFN-beta (ELISA) induced by LPS and by PAM3CSK4 plus baseline cytokine levels (no exposure to LPS or PAM3CSK4). Urinary levels of protein will be quantified in some studies as a measure of early kidney dysfunction.

We hope the results of this study may lead to discovery of important information regarding the role of MDC1 (Mediator of DNA damage Checkpoint protein 1) in human disease, potentially identifying new targets for future studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female 18 years of age or older
* Participants must be able to understand and provide written informed consent to participate in the study
* Participants must be able to travel to the CRU
* Willing and able to fast after midnight the night prior to their study appointment
* Healthy participants as defined by the International Red Cross guidelines (Healthy means that an individual feels well and can perform normal activities. If the individual has a chronic condition such as diabetes or high blood pressure, healthy also means that they are being treated and the condition is under control).

EXCLUSION CRITERIA:

* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within 5 days prior to enrollment visit (e.g., Motrin, ibuprofen, naproxen, and Advil)
* Use of acetaminophen (Tylenol) within 5 days prior to enrollment visit
* Use of cholesterol lowering drugs (statins) within 30 days prior to enrollment visit (e.g., Zocor, Mevacor, Lipitor, and Crestor)
* Use of immunosuppressants or other immune-modifying drugs [e.g., Rituxan, Humira, Enbrel, Cyclosporin (Neoral, Sandimmune, and SangCya), and Azathioprine (Imuran)], Monoclonal antibodies [e.g., infliximab (Remicade)], and corticosteroids (e.g., prednisone, prednisolone and dexamethasone)
* Current treatment for cancer with chemotherapy or radiation
* Confirmed or suspected immunosuppressive or immunodeficient condition
* GI or respiratory Illness within 5 days prior to enrollment visit, including cold or allergies
* Smoked tobacco, chewed tobacco or used electronic cigarettes within 2 weeks prior to enrollment visit (for participants who provide a urine specimen, this will be defined by urine cotinine >200 ng/mL at visit)
* Alcohol consumption greater than 2 standard drinks (1 standard drink contains 15 g of ethanol) per day within the last 24 hours prior to the enrollment visit
* Body weight < 50 kg (<110 lbs)
* Temperature > 37.6 C; blood pressure < 90/50 mm Hg or > 170/95 mm Hg; pulse rate < 50 or >100 beats/minute
* Pregnant or suspected pregnancy
* Chronic Kidney Disease

The PI may review medication use on a case by case basis and make a medical determination on the participant s eligibility. In these cases, the PI determination will be documented in the participant s chart.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in Environmental Polymorphism Registry (EPR)@@@
Sampling Method: Non-Probability Sample
Enrollment: 725 (Estimated)
Dates: Start 2012-07-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of this study are for both cell types and will be levels of 6 cytokines [TNF alpha, IL-6, MIP-2, IL-8, MCP-1, and IFN-beta (ELISA)] induced by LPS and by PAM3CSK4 plus baseline cytokine levels (no exposure to LPS or PAM3CSK... | After analysis
  The primary endpoints of this study are for both cell types and will be levels of 6 cytokines [TNF alpha, IL-6, MIP-2, IL-8, MCP-1, and IFN-beta (ELISA)] induced by LPS and by PAM3CSK4 plus baseline cytokine levels (no exposure to LPS or PAM3CSK4).

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Fessler, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
It isn t known yet if there will be a plan to make IPD available

REFERENCES:
- [Background] Castiblanco J, Varela DC, Castano-Rodriguez N, Rojas-Villarraga A, Hincapie ME, Anaya JM. TIRAP (MAL) S180L polymorphism is a common protective factor against developing tuberculosis and systemic lupus erythematosus. Infect Genet Evol. 2008 Sep;8(5):541-4. doi: 10.1016/j.meegid.2008.03.001. Epub 2008 Mar 12. PMID 18417424
- [Background] Singaraja RR, Brunham LR, Visscher H, Kastelein JJ, Hayden MR. Efflux and atherosclerosis: the clinical and biochemical impact of variations in the ABCA1 gene. Arterioscler Thromb Vasc Biol. 2003 Aug 1;23(8):1322-32. doi: 10.1161/01.ATV.0000078520.89539.77. Epub 2003 May 22. PMID 12763760
- [Background] Kenny EF, O'Neill LA. Signalling adaptors used by Toll-like receptors: an update. Cytokine. 2008 Sep;43(3):342-9. doi: 10.1016/j.cyto.2008.07.010. Epub 2008 Aug 15. PMID 18706831
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-E-0129.html